CLINICAL TRIAL: NCT02284191
Title: The Role of Early CT Coronary Angiography in the Evaluation, Intervention and Outcome of Patients Presenting to the Emergency Department With Suspected or Confirmed Acute Coronary Syndrome.
Brief Title: Rapid Assessment of Potential Ischaemic Heart Disease With CTCA
Acronym: RAPID-CTCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RAPID-CTCA-2014
Record Dates: First submitted 2014-10-06; First posted 2014-11-05 (Estimated); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Radiology; Acute Medicine; Emergency Medicine; Cardiology
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT Coronary Angiogram (Active Comparator): CT Coronary Angiogram plus standard care
  Interventions: Radiation: CT Coronary Angiogram
- Standard Care (No Intervention): Standard care only

INTERVENTIONS:
Radiation: CT Coronary Angiogram — Completion of a CT Coronary Angiogram
  Arms: CT Coronary Angiogram

SUMMARY:
This study aims to investigate the effect of early CTCA in patients with suspected or confirmed Acute Coronary Syndrome (ACS) presenting to the Emergency Department (ED) or Medical Assessment Unit (MAU), upon interventions, event rates and health care costs in a pragmatic clinical trial and economic evaluation up to 1 year after the trial intervention. The primary objective will be to investigate the effect of the intervention on all-cause death or subsequent type 1 or type 4b MI at one year, measured as time to first such event.

DETAILED DESCRIPTION:
DESIGN: Open parallel group randomised controlled trial of early computed tomography coronary angiography (CTCA) in patients presenting with suspected/confirmed acute coronary syndrome (ACS) to Emergency Departments (ED) and Medical Assessment Units.

SETTING: 37 EDs, radiology, cardiology and acute medical services in tertiary/district general National Health Service (NHS) hospitals.

TARGET POPULATION: Inclusion Criteria: Patient ≥18 years with symptoms mandating investigation for suspected or confirmed ACS with at least one of: ECG abnormalities e.g. ST segment depression >0.5 mm; History of ischaemic heart disease (where the clinician assessing patient confirms history based on patient history or available records); Troponin elevation above the 99th centile of the normal reference range or increase in high sensitivity troponin meeting European Society of Cardiology criteria for 'rule-in' or myocardial infarction (NB troponin assays will vary from site to site; local laboratory reference standards will be used). Exclusion Criteria: 1.Signs, symptoms, or investigations supporting high-risk ACS: ST elevation MI; ACS with signs or symptoms of acute heart failure or circulatory shock; Crescendo episodes of typical anginal pain; Marked or dynamic ECG changes e.g. ST depression of >3 mm; Clinical team have scheduled early invasive coronary angiography on day of trial eligibility assessment. 2. Patient inability to undergo CT: Severe renal failure (serum creatinine >250 µmol/L or estimated glomerular filtration rate <30 mL/min); Contrast allergy; Beta blocker intolerance (if no alternative heart rate limiting agent available/suitable) or allergy; Inability to breath hold; Atrial fibrillation (where mean heart rate is anticipated to be greater than 75 beats per minute after beta blockade). 3. Patient has had invasive coronary angiography or CTCA within last 2 years and the previous investigation revealed obstructive coronary artery disease, or patient had either investigation within the last 5 years and the result was normal. 4.Previous recruitment to the trial; 5.Known pregnancy or currently breast feeding; 6. Inability to consent; 7.Further investigation for ACS would not in the patient's interest, due to limited life expectancy, quality of life or functional status; 8.Prisoners

HEALTH TECHNOLOGIES BEING ASSESSED: Early use of ≥64-slice CTCA as part of routine assessment compared to standard care.

MEASUREMENT OF COSTS/OUTCOMES: Primary end-point will be one-year all-cause death or subsequent type 1 or type 4b MI at one year, measured as time to first such event. Secondary endpoints: Key Secondary Endpoints : 1. Coronary Heart Disease (CHD) death or subsequent non-fatal MI; 2. Cardiovascular Disease (CVD) death or subsequent non-fatal MI; 3. Subsequent non-fatal MI; 4.Coronary Heart Disease death; 5. Cardiovascular death; 6. All-cause death. Other Endpoints; Coronary

Heart Disease (CHD) death or subsequent non-fatal MI (type 1 or 4b);Subsequent Non-fatal MI (type 1 or 4b); Non-cardiovascular death; Invasive coronary angiography; Coronary revascularisation; Percutaneous coronary intervention; Coronary artery bypass graft; Proportion of patients prescribed ACS therapies during index hospitalisation; Proportion of patients discharged on preventative treatment or have alteration in dosage of preventative treatment during index hospitalisation; Length of stay for index hospitalisation; Representation or rehospitalisation with suspected ACS/recurrent chest pain within 12 months after index hospitalisation; Chest pain symptoms up to 12 months; Patient satisfaction at 1 month; Clinician certainty of presenting diagnosis after CTCA; Quality of Life (measured by EQ- 5D-5L up to12 months). Adverse Events and Serious Adverse Events; Proportion of patients with alternative cardiovascular diagnoses identified on CTCA; Proportion of patients with non-cardiovascular diagnosis identified on CTCA; Radiation exposure from CTCA as trial intervention. Cost effectiveness:

Estimated in terms of the lifetime incremental cost per quality-adjusted life year (QALY) gained.

SAMPLE SIZE: 1,749 patients (1,748 available for analysis).

ELIGIBILITY:
INCLUSION CRITERIA

Patient ≥18 years with symptoms mandating investigation for suspected or confirmed ACS with at least one of:

* ECG abnormalities e.g. ST segment depression >0.5 mm;
* History of ischaemic heart disease (where the clinician assessing patient confirms history based on patient history or available records);
* Troponin elevation above the 99th centile of the normal reference range or increase in high sensitivity troponin meeting European Society of Cardiology criteria for 'rule-in' or myocardial infarction (NB troponin assays will vary from site to site; local laboratory reference standards will be used).

EXCLUSION CRITERIA

* Signs, symptoms, or investigations supporting high-risk ACS:

  * ST elevation MI;
  * ACS with signs or symptoms of acute heart failure or circulatory shock;
  * Crescendo episodes of typical anginal pain;
  * Marked or dynamic ECG changes e.g. ST depression of >3 mm
  * Clinical team have scheduled early invasive coronary angiography on day of trial eligibility assessment.
* Patient inability to undergo CT:

  * Severe renal failure (serum creatinine >250 µmol/L or estimated glomerular filtration rate <30 mL/min);
  * Contrast allergy;
  * Beta blocker intolerance (if no alternative heart rate limiting agent available/suitable) or allergy ;
  * Inability to breath hold;
  * Atrial fibrillation (where mean heart rate is anticipated to be greater than 75 beats per minute after beta blockade).
* Patient has had invasive coronary angiography or CTCA within last 2 years and the previous investigation revealed obstructive coronary artery disease, or patient had either investigation within the last 5 years and the result was normal.
* Previous recruitment to the trial;
* Known pregnancy or currently breast feeding;
* Inability to consent;
* Further investigation for ACS would not in the patient's interest, due to limited life expectancy, quality of life or functional status;
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1749 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair J Gray, Principal Investigator — NHS Lothian
Locations (37):
- Jersey General Hospital, Saint Helier, Jersey
- United Kingdom (36):
  - Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon
  - Ulster Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - The Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Russells Hall Hospital, Dudley
  - Ninewells Hospital, Dundee
  - Royal Infirmary Edinburgh, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Raigmore Hospital, Inverness
  - Victoria Hospital, Kirkcaldy
  - Leeds General Infirmary, Leeds
  - University Hospital Lewisham, Lewisham
  - Royal London Hospital, London
  - St. Thomas' Hospital, London
  - University Hospital North Tees, London
  - Whipps Cross Hospital, London
  - Luton & Dunstable Hospital, Luton
  - Borders General Hospital, Melrose
  - Milton Keynes University Hospital NHS Foundation Trust, Milton Keynes
  - Royal Victoria Infirmary, Newcastle
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire NHS Foundation Trust, Reading
  - East Surrey Hospital, Redhill
  - Rotherham Hospital, Rotherham
  - Sandwell General Hospital, Sandwell
  - Northern General Hospital, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - University Hospitals of the Midlands, Stoke
  - Torbay Hospital, Torquay
  - New Cross Hospital, Wolverhampton
  - Worcestershire Royal Hospital, Worcester
  - Wrexham Maelor Hospital, Wrexham
  - University Hospital South Manchester, Wythenshawe

REFERENCES:
- [Result] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Derived] Lakshmanan S, Wang KL, Meah MN, Tzolos E, Bularga A, Dweck MR, Curzen N, Kardos A, Keating L, Storey RF, Mills NL, Slomka PJ, Dey D, Gray A, Williams MC, Roobottom C, Newby DE. Diagnostic and Prognostic Performance of Pericoronary Adipose Tissue Attenuation in Suspected Acute Coronary Syndrome: Insights from the RAPID-CTCA Trial. Radiol Cardiothorac Imaging. 2026 Feb;8(1):e250074. doi: 10.1148/ryct.250074. PMID 41504639
- [Derived] Wang KL, Taggart C, McDermott M, O'Brien R, Oatey K, Keating L, Storey RF, Felmeden D, Curzen N, Kardos A, Roobottom C, Smith J, Goodacre S, Newby DE, Gray AJ; RAPID-CTCA Investigators. Clinical decision aids and computed tomography coronary angiography in patients with suspected acute coronary syndrome. Emerg Med J. 2024 Jul 22;41(8):488-494. doi: 10.1136/emermed-2024-213904. PMID 38857986
- [Derived] Meah MN, Tzolos E, Wang KL, Bularga A, Dweck MR, Curzen N, Kardos A, Keating L, Storey RF, Mills NL, Slomka PJ, Dey D, Newby DE, Gray A, Williams MC, Roobottom C. Plaque Burden and 1-Year Outcomes in Acute Chest Pain: Results From the Multicenter RAPID-CTCA Trial. JACC Cardiovasc Imaging. 2022 Nov;15(11):1916-1925. doi: 10.1016/j.jcmg.2022.04.024. Epub 2022 Jun 15. PMID 36357133
- [Derived] Meah MN, Bularga A, Tzolos E, Chapman AR, Daghem M, Hung JD, Chiong J, Taggart C, Wereski R, Gray A, Dweck MR, Roobottom C, Curzen N, Kardos A, Felmeden D, Mills NL, Slomka PJ, Newby DE, Dey D, Williams MC. Distinguishing Type 1 from Type 2 Myocardial Infarction by Using CT Coronary Angiography. Radiol Cardiothorac Imaging. 2022 Oct 27;4(5):e220081. doi: 10.1148/ryct.220081. eCollection 2022 Oct. PMID 36339063
- [Derived] Gray AJ, Roobottom C, Smith JE, Goodacre S, Oatey K, O'Brien R, Storey RF, Curzen N, Keating L, Kardos A, Felmeden D, Lee RJ, Thokala P, Lewis SC, Newby DE. Early computed tomography coronary angiography in adults presenting with suspected acute coronary syndrome: the RAPID-CTCA RCT. Health Technol Assess. 2022 Aug;26(37):1-114. doi: 10.3310/IRWI5180. PMID 36062819
- [Derived] Gray AJ, Roobottom C, Smith JE, Goodacre S, Oatey K, O'Brien R, Storey RF, Curzen N, Keating L, Kardos A, Felmeden D, Lee RJ, Thokala P, Lewis SC, Newby DE; RAPID-CTCA Investigators. Early computed tomography coronary angiography in patients with suspected acute coronary syndrome: randomised controlled trial. BMJ. 2021 Sep 29;374:n2106. doi: 10.1136/bmj.n2106. PMID 34588162
- [Derived] Gray AJ, Roobottom C, Smith JE, Goodacre S, Oatey K, O'Brien R, Storey RF, Na L, Lewis SC, Thokala P, Newby DE. The RAPID-CTCA trial (Rapid Assessment of Potential Ischaemic Heart Disease with CTCA) - a multicentre parallel-group randomised trial to compare early computerised tomography coronary angiography versus standard care in patients presenting with suspected or confirmed acute coronary syndrome: study protocol for a randomised controlled trial. Trials. 2016 Dec 7;17(1):579. doi: 10.1186/s13063-016-1717-2. PMID 27923390
- See also: Protocol publication — https://www.ncbi.nlm.nih.gov/pubmed/27923390
- See also: Final Publication — https://www.bmj.com/content/374/bmj.n2106.full
- See also: Lay Summary of Results — https://www.ed.ac.uk/usher/edinburgh-clinical-trials/our-studies/completed-studies/rapid-ctca
- See also: Lay Summary of Results — https://www.emergeresearch.org/trial/rapid-ctca/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1749 participants were enrolled into the study but only 1748 were available for analysis due to one participant requesting all their data be withdrawn from the dataset. Their randomisation allocation is unknown.
Groups:
- CTCA Plus Standard Care: Computed tomography coronary angiogram plus standard care
Period: Overall Study
Arm/Group | CTCA Plus Standard Care | Standard Care
Started | 877 | 871
Completed | 875 | 868
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT Coronary Angiogram | Standard Care | Total
Number analyzed (Participants) | 877 | 871 | 1748
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 502 | 517 | 1019
  >=65 years | 375 | 354 | 729
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (12.2) | 61.2 (13.0) | 61.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 313 | 321 | 634
  Male | 564 | 550 | 1114
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 858 | 851 | 1709
  Jersey | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: All-cause Death or Subsequent Non-fatal Type 1 or Type 4b MI at One Year Measured as Time to First Such Event.
Description: Number of participants categorised as having primary outcome event - all-cause death or subsequent non-fatal myocardial infarction (type 1 or 4b) at one year (post randomisation), measured as time to first such event. Myocardial infarction 'type' was defined according to the most recent Universal Definition (1). and was adjudicated independently by two cardiologists blinded to the intervention and the categorisation added to the study database.
Time Frame: 1 year (post randomisation)
Population: All randomised participants
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 51 | 53

2. Secondary Outcome: Coronary Heart Disease Death or Subsequent Non-fatal MI
Description: Number of participants with coronary heart disease death or subsequent non-fatal myocardial infarction, one year after randomisation.
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 47 | 45

3. Secondary Outcome: Cardiovascular Disease Death or Subsequent Non-fatal MI
Description: Number of participants categorised as having cardiovascular disease death or subsequent non-fatal myocardial infarction, one year after randomisation
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 48 | 46

4. Secondary Outcome: Subsequent Non-fatal MI
Description: Number of participants with subsequent non-fatal myocardial infarction, at one year post-randomisation.
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 39 | 40

5. Secondary Outcome: Coronary Heart Disease Death
Description: Number of participants with Coronary Heart Disease deaths, one year after randomisation
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 11 | 6

6. Secondary Outcome: Cardiovascular Death
Description: Number of participants with cardiovascular death, one year after randomisation
Time Frame: 1 year (post-randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 12 | 8

7. Secondary Outcome: All-cause Death
Description: Number of participants with "all-cause" death, one year post-randomisation
Time Frame: 1 year (post-randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 19 | 17

8. Secondary Outcome: Coronary Heart Disease (CHD) Death or Subsequent Non-fatal MI (Type 1 or 4b)
Description: Number of participants with Coronary heart disease death or subsequent non-fatal myocardial infarction (type 1 or 4b), one year after randomisation
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 43 | 43

9. Secondary Outcome: Subsequent Non-fatal MI (Type 1 or 4b)
Description: Number of participants with subsequent non-fatal myocardial infarction (type 1 or 4b), one year post randomisation
Time Frame: 1 year (post-randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 35 | 38

10. Secondary Outcome: Non-cardiovascular Death
Description: Number of participants with non-cardiovascular deaths, one year post-randomisation
Time Frame: 1 year (post-randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 7 | 9

11. Secondary Outcome: Invasive Coronary Angiography
Description: Number of participants with Invasive coronary angiography procedures, one year post-randomisation
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 474 | 530

12. Secondary Outcome: Coronary Revascularisation
Description: Number of participants with Coronary revascularisation by percutaneous coronary intervention or coronary artery bypass graft surgery, one year post randomisation
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 300 | 288

13. Secondary Outcome: Percutaneous Coronary Intervention
Description: Number of participants with percutaneous coronary interventions, 1 year (post randomisation)
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 260 | 240

14. Secondary Outcome: Coronary Artery Bypass Graft
Description: Number of participants with coronary artery bypass graft procedures, 1 year post randomisation
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 52 | 55

15. Secondary Outcome: Number of Patients Prescribed ACS Therapies During Index Hospitalisation
Description: Number of participants prescribed acute coronary syndrome therapies during index hospitalisation, 1 year (post randomisation)
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 595 | 580

16. Secondary Outcome: Discharged on Preventative Treatment or Alteration in Dosage of Preventative Treatment During Index Hospitalisation
Description: Number of participants discharged on preventative treatment having not been on preventative treatment prior to index hospitalisation, or alteration of dosage of preventative treatment during index hospitalisation, i.e. change in prevention treatment during index hospitalisation.
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 554 | 539

17. Secondary Outcome: Length of Stay for Index Hospitalisation
Description: Length of Stay for Index Hospitalisation visit, measured in days each participants was hospitalised prior to their discharge. There is no maximum length an index hospitalisation might be for an individual participant, but follow up of participants is for a maximum one year.
Time Frame: A maximum follow up of one-year post-randomisation.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
days | 2.2 [1.1 to 4.1] | 2.0 [1.0 to 3.8]

18. Secondary Outcome: Representation or Rehospitalisation With Suspected ACS/ Recurrent Chest Pain After Index Hospitalisation
Description: Number of participants who represented or were rehospitalised with suspected acute coronary syndrome/recurrent chest pain after discharge from index hospitalisation, up to one year after randomisation
Time Frame: 1 year (post randomisation)
Measure: Count of Participants; unit: Participants
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 877 | 871
Participants | 138 | 130

19. Secondary Outcome: Radiation Exposure From CTCA as Trial Intervention
Description: Median effective radiation dose (mSv) from CTCA received by participants in the CTCA arm of the study. Value derived from dose length product (mGy/cm) using conversion factor of 0.014 mSv/mGy/cm.
Time Frame: 1 year (post randomisation)
Population: Standard care group do not get CT so there is no data to analyse
Measure: Median (Inter-Quartile Range); unit: mSv
Arm/Group | CT Coronary Angiogram | Standard Care
Number analyzed (Participants) | 767 | 0
mSv | 3.1 [1.9 to 5.5] |

ADVERSE EVENTS:
Time Frame: Protocol defined adverse events were recorded/reported from consent until 10 days after joining the study. Anticipated events which formed the study outcomes (e.g -death, MI) were recorded for one year post randomisation. No other events were recorded
Description: Serious Adverse Events related to endpoints collected and reported. Protocol defined AEs collected only: Contrast related anaphylaxis/allergy requiring treatment, critical care admission or resulting in cardiac arrest/ death, Contrast related AKI or Acute on CKD, Side effects related to beta blocker, HR-limiting medication or GTN.
Arm/Group | CT Coronary Angiogram | Standard Care
All-Cause Mortality (participants affected / at risk) | 19/877 | 17/871
Serious Adverse Events (participants affected / at risk) | 18/877 | 10/871
Other Adverse Events (participants affected / at risk) | 3/877 | 0/871
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT Coronary Angiogram (N=877) | Standard Care (N=871)
Readmission with non-cardiac condition (General disorders) | 6 (6) | 2 (2)
Readmission with chest pain - not CHD related (General disorders) | 2 (2) | 4 (4)
Readmission with chest pain - CHD related (General disorders) | 3 (3) | 2 (2)
Readmission with chest pain - unclear (General disorders) | 1 (1) | 2 (2)
Not related - other (General disorders) | 5 (5) | 0 (0) — Not related/relevant to trial intervention/research question
Patient deterioration prior to CTCA (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT Coronary Angiogram (N=877) | Standard Care (N=871)
IV cannula issue (Surgical and medical procedures) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT02284191/Prot_001.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02284191/SAP_000.pdf